CLINICAL TRIAL: NCT02225080
Title: Duragen® Secure Post Marketing Clinical Follow-up (PMCF)
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: N-DURSEC-001
Record Dates: First submitted 2014-07-28; First posted 2014-08-25 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Dura Mater Nick Cut or Tear; Surgery
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Duragen Secure: Have undergone a neurosurgical procedure where DuraGen® Secure has been implanted

SUMMARY:
The purpose of this study is to gather information about post-market performance of DuraGen Secure.The aim of this post market clinical follow-up (PMCF) is to obtain post market clinical data to evaluate the presence of unintended residual risks associated with the use of DuraGen Secure that were not anticipated or identified in the animal studies, bench studies or clinical evaluation report.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have undergone a neurosurgical procedure where DuraGen® Secure has been implanted

Exclusion Criteria:

* Patient who does not agree to allow collection of his/her medical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurgosurgery service in Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Hopital Lariboisière, Paris, France
- die Charité - Universitätsmedizin Berlin, Berlin, Germany
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe, Valencia
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duragen Secure
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Duragen Secure
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient's Outcome
Description: Patient outcome from the procedure (recovered without sequelae, ongoing with medical intervention, ongoing with surgical intervention, deceased, other)
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Duragen Secure
Number analyzed (Participants) | 100
Participants
  Recovered without sequelae | 73
  Ongoing with medical intervention | 7
  Ongoing with surgical intervention | 15
  Deceased | 3
  Other | 2

2. Secondary Outcome: Occurence of Adverse Event
Description: Adverse event that occured 72 hours post-operatively
Time Frame: first 72 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Duragen Secure
Number analyzed (Participants) | 100
Participants | 19

3. Secondary Outcome: Occurence of Adverse Event
Description: Adverse event that occured between days 4-14 post-operatively
Time Frame: between days 4-14
Measure: Count of Participants; unit: Participants
Arm/Group | Duragen Secure
Number analyzed (Participants) | 100
Participants | 18

4. Secondary Outcome: Occurence of Adverse Event
Description: Adverse event that occured between days 15-30 post-operatively
Time Frame: Between days 15-30
Measure: Count of Participants; unit: Participants
Arm/Group | Duragen Secure
Number analyzed (Participants) | 100
Participants | 15

ADVERSE EVENTS:
Time Frame: Retrospective chart review of AE occured between surgery (Day 0) and file completion (between Day 30 and Day 60)
Arm/Group | Duragen Secure
All-Cause Mortality (participants affected / at risk) | 3/100
Serious Adverse Events (participants affected / at risk) | 31/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duragen Secure (N=100)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrhythmia (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Inflammatory reaction (General disorders) | 3
Wound healing disturbance (General disorders) | 1
Death (General disorders) | 2
Weakness worsened (General disorders) | 1
Infection (Infections and infestations) | 4
Meningitis (Infections and infestations) | 5
subdural empyema (Infections and infestations) | 1
Shunt infection (Infections and infestations) | 1
cerebral empyema (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Anemia postoperative (Injury, poisoning and procedural complications) | 1
Postoperative bleeding (Injury, poisoning and procedural complications) | 1
Graft failure (Injury, poisoning and procedural complications) | 1
Cardiac enzymes increased (Investigations) | 1
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CSF leakage (Nervous system disorders) | 2
Haematoma cerebral (Nervous system disorders) | 1
Intracranial haemorrhage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Subdural Hygroma (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 3
Paraparesis (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 2
Hemorrhage intracranial (Nervous system disorders) | 1
Intracranial hypertension (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 3
Organic brain syndrome (Psychiatric disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Brain tumor operation (Surgical and medical procedures) | 1
Thrombosis venous deep (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less